CLINICAL TRIAL: NCT05290129
Title: Oxytocin Maintenance Infusion in Labouring Women Undergoing Cesarean Delivery: an Up-down Sequential Allocation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-02
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Hemorrhage
Keywords: Cesarean delivery; oxytocin; uterotonic; pregnancy; labour
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Biased coin up-and-down design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Oxytocin infusion rate 4 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 4 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 6 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 6 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 10 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 10 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 14 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 14 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 18 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 18 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 22 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 22 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 26 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 26 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 30 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 30 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 34 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 34 IU/h.
  Interventions: Drug: Oxytocin
- Oxytocin infusion rate 36 IU/h (Experimental): The maintenance infusion rate of oxytocin will be 36 IU/h.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin will be prepared in a 1L bag of Ringer's lactate, to be infused at a rate of 125 ml/h.
  Other Names: Pitocin

SUMMARY:
This study is designed to determine the minimal effective oxytocin maintenance infusion required in labouring women undergoing cesarean delivery to achieve the best effect. Oxytocin is a drug that is routinely used to help the uterus to contract and keep it contracted after delivery. Consequently, it will help to reduce blood loss after delivery. In order to determine the minimal effective dose, the investigators will conduct a dose-finding study. The first patient will receive a set oxytocin infusion. The next patient's infusion dose of oxytocin, will either increase or decrease, depending on how the previous patient responds in terms of uterine tone. If the response is satisfactory with the infusion dose used, the next patient will either receive the same infusion dose or it will be decreased depending on a probability of 1:9. If the response is not satisfactory, then the infusion dose will increase for the next patient. The dose for each patient will be determined based on the results of the uterine contraction of the previous patient.

The investigators hypothesize that the ED90 of the oxytocin infusion rate to maintain adequate uterine tone in labouring women with induced or augmented labour undergoing cesarean delivery, following an initial effective bolus dose, would be lower than 0.74 IU/min (44 IU/h), which was found as the ED90 in a previous study, without an initial bolus dose prior to the infusion.

DETAILED DESCRIPTION:
This study will be conducted as a prospective, double blinded clinical trial (patient, anesthesiologist and obstetrician blinded to the oxytocin dose), in an up-down sequential allocation fashion. The objective of the study is to determine the minimum effective dose of oxytocin infusion required to produce appropriate uterine contraction during and after cesarean delivery under neuraxial anesthesia in laboring women. For the purpose of this study, the minimum effective dose is defined to be that at which adequate response occurs in 90% of patients, i.e. ED90.

ELIGIBILITY:
Inclusion Criteria:

• All patients with induced or augmented labour undergoing cesarean delivery under neuraxial anesthesia (at least 3 hours of prior exposure to oxytocin during labour)

Exclusion Criteria:

* All patients who refuse to give written informed consent
* All patients who declare allergy or hypersensitivity to oxytocin
* A history of hypertension and/or severe cardiac disease(s)
* All patients who have contraindications for neuraxial anesthesia
* All patients who will be converted to general anesthesia intraoperatively
* All patients with placenta previa and multiple gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Uterine tone up to discharge from the post anesthetic care unit (PACU): questionnaire | 2 hours
  Uterine tone will be evaluated as satisfactory or unsatisfactory by the obstetrician throughout the surgery, starting at 5 minutes after the oxytocin infusion. It will also be measured at 10 minutes following the oxytocin infusion and every 10 minutes following that for the duration of the surgery. Unsatisfactory uterine tone at any time until discharge from the PACU will be considered a failure of the maintenance infusion.

SECONDARY OUTCOMES:
Calculated blood loss | 24 hours
  Estimated blood loss will be calculated using the difference in hematocrit values prior to surgery and 24 hours post surgery, using the following formula:
  Calculated blood loss (mL) = EBV ((Pre-op Htc-Post-op Htc)/pre-op Htc) EBV (estimated blood volume) in ml: patient's weight in kg x 85.
Need for blood transfusion | 24 hours
  Blood product administered.
Episodes of bleeding postpartum | 24 hours
  Number of episodes of bleeding postpartum up to 24 hours post delivery.
Intraoperative requirement for additional uterotonic medication | 1 hour
  A request made by the obstetrician performing the cesarean delivery for additional uterotonic medication, due to bleeding or poor uterine tone.
Requirement for additional uterotonic medication in the PACU | 2 hours
  Any uterotonic medication administered while the patient is in PACU
Requirement for additional uterotonic medication from discharge from the PACU until 24 hours postpartum. | 24 hours
  Any uterotonic medication administered after the patient is discharged from PACU until 24 hours postpartum.
Hypotension: systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, from drug administration until end of surgery
Hypertension: systolic blood pressure greater than 120% of baseline | 2 hours
  Systolic blood pressure > 120% of baseline, from drug administration until end of surgery
Tachycardia: heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, from drug administration until end of surgery
Bradycardia: heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline or a heart rate < 50bpm, from drug administration until end of surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, from drug administration until end of surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, from drug administration until end of surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, from drug administration until end of surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea and number of episodes, from drug administration until end of surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting and number of episodes, from drug administration until end of surgery
Presence of chest pain: questionnaire | 2 hours
  Any presence of chest pain, from drug administration until end of surgery, as reported by the patient
Presence of shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, from drug administration until end of surgery, as reported by the patient
Presence of headache: questionnaire | 2 hours
  Any presence of headache, from drug administration until end of surgery, as reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No